CLINICAL TRIAL: NCT05195606
Title: The Effect of Auditory and Tactile Stimulus on Consciousness, Oxygen Saturation, and Mean Arterial Pressure in Traumatic Coma Patients: A Randomized Controlled Single-Blind Study
Brief Title: The Effect of Auditory and Tactile Stimuli in Traumatic Coma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Arş. Gör. Arzu TAT ÇATAL, Principal Investigator, Akdeniz University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: KAEK-724
Record Dates: First submitted 2021-12-29; First posted 2022-01-19 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Head Trauma; Traumatic Coma; Nursing Caries
Keywords: Head trauma; Nursing; Auditory stimulus; Tactile stimulus; Foot massage; Consciousness; Coma
MeSH Terms: conditions — Craniocerebral Trauma; Coma, Post-Head Injury; Coma

STUDY DESIGN:
Who Masked: Participant
Masking Description: In the application process, single blinding will be provided as the patients do not know which group they are included in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (No Intervention): There is no standard sensory stimulation program for comatose patients with head trauma in the hospitals where the research will be conducted. Therefore, the control group will receive routine practice.
- Auditory stimulus (Intervention A) (Experimental): Auditory stimulus for patients in this group
  Interventions: Other: Auditory stimulus
- Tactile stimulus (Intervention B) (Experimental): Tactile stimulus for patients in this group
  Interventions: Other: Tactile stimulus

INTERVENTIONS:
Other: Auditory stimulus — Auditory stimulus will be applied to the patients in intervention group A. For the auditory stimulus, the sound recording of the relatives of the patients will be taken and the patients will be listened to with headphones.
  Arms: Auditory stimulus (Intervention A)
Other: Tactile stimulus — Tactile stimulus will be applied to the patients in the intervention group B. The tactile stimulus will be performed by the researcher with a foot massage to be applied to the patient.
  Arms: Tactile stimulus (Intervention B)

SUMMARY:
This study focused on examining the effects of auditory and tactile stimuli to reduce sensory deprivation on consciousness, oxygen saturation and mean arterial pressure in traumatic coma patients.

DETAILED DESCRIPTION:
Background: One of the most important problems experienced by patients treated in the intensive care unit due to traumatic coma is sensory deprivation.

Aim: In this study, it was aimed to examine the effects of auditory and tactile stimulus to be used in the prevention of sensory deprivation on consciousness, oxygen saturation and mean arterial pressure.

Study Design: The study was planned as a randomized controlled single-blind experiment with three groups. In the study, the patients in the Control group will be given a routine application, the patients in the Intervention A group will be given auditory stimuli, and the patients in the Intervention B group will be treated with tactile stimulus. Interventions will be administered once a day for seven days, for a total of seven times. The "block randomization method" was chosen as the randomization method. In this study, hospitals were taken as a block. An equal number of patients will be recruited from two hospitals and 15 patients will be distributed to three groups from each hospital using the "simple randomization method". 30 patients in each group and 90 patients in total will be included in the study.

Methods: The researcher applied to the patients hospitalized in the intensive care unit for 24-72 hours for seven days, once a day (seven times in total) between 10:00 and 15:00 (Intervention A: 10 minutes of audio recording will be played with headphones. Intervention B: 10 minutes) (5 minutes for one foot) foot massage will be applied. Glaskow Coma Score, oxygen saturation and Mean Arterial Pressure will be measured before and after each intervention (twice daily).

ELIGIBILITY:
Inclusion Criteria:

* Being treated in the intensive care unit for at least 24 hours due to traumatic coma,
* 18 years and older
* Relatives of those who agreed to participate in the study
* GCS score between 3-8 (GCS: 3-8 indicates coma)
* Without hearing impairment
* Having no authority for auditory stimulus
* No problem for foot massage (Lower extremity fracture, infection)

Exclusion Criteria:

* Who are under the age of 18
* Those whose relatives do not agree to participate in the research
* GKS score above 8

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-06-15 (Estimated); Primary Completion 2024-10-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Glasgow Coma Scale (GCS) | 1 week
  GCS is a diagnostic tool that provides objective evaluation of the patient's eye-opening, verbal and motor response to stimuli. In the scale, the eye opening score is between 1-4, the verbal response is between 1-5, and the motor response is between 1-6, and the total score is between 3-15. The GCS score of the patient who did not respond to painful stimuli, could not open his eyes spontaneously, and had complete loss of muscular tone was three; The GCS score of the patient who is oriented, spontaneously opens his eyes and fulfills the orders is 15. It should be understood that the patient with a GCS score of less than eight is in a coma.